CLINICAL TRIAL: NCT00802776
Title: Comparison of Femtosecond Laser-Assisted and Traditional Keratoplasty for Keratoconus
Brief Title: Femtosecond Laser Assisted Keratoplasty
Acronym: FLAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shahzad Mian, erry J Bergstrom Collegiate Professor of Resident Education in Ophthalmology and Visual Sciences and Associate Professor of Oph, Ophthalmology & Visual Science, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM 15615-FLAK
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLAK (Active Comparator): Femtosecond laser assisted keratoplasty
  Interventions: Procedure: Femtosecond laser assisted keratoplasty
- PKP (Active Comparator): Penetrating Keratoplasty
  Interventions: Procedure: PKP

INTERVENTIONS:
Procedure: Femtosecond laser assisted keratoplasty
  Arms: FLAK
Procedure: PKP
  Arms: PKP

SUMMARY:
Penetrating keratoplasty (PKP) is corneal transplantation performed by using round trephine blades to create matched circumferential incisions in both the diseased cornea and the donor cornea. The donor tissue graft is then secured in place with sutures which are usually removed postoperatively.The primary surgical goals are the preservation of a clear graft and improvement of vision. Surgical outcomes are limited by donor-recipient junction mismatch, astigmatism, rejection, infection and wound dehiscence.

The femtosecond laser is a focusable, infrared laser capable of cutting tissue at various depths and in a range of patterns, and is currently being used to create corneal lamellar flaps in LASIK surgery. The laser parameters can be adjusted for submicron precision in cutting desired diameters, depths and shapes in the cornea, with minimal collateral injury. This technology is now capable of creating full-thickness corneal trephinations with customized locking edges at the graft-host junction between the donor and recipient corneas in Femtosecond Laser-Assisted Keratoplasty (FLAK). This approach may allow for better wound junction of the donor and recipient corneas, which in turn may also significantly reduce astigmatism, improve wound healing and visual recovery.

This pilot study will help us determine optimal femtosecond laser spot size, separation, fluence, and energy which result in the best graft-host fit.

The specific aim is to investigate postoperative physiology and biomechanics after FLAK in human eyes.

DETAILED DESCRIPTION:
Penetrating keratoplasty (PKP) or full-thickness corneal transplantation is a common and highly successful method to restore vision decreased by corneal opacification. Surgery is performed by using round trephine blades to create matched circumferential incisions in both the diseased cornea and the donor cornea. Several types of blades are currently available to create uniform corneal cuts. The donor tissue graft is then secured in place with sutures which are usually removed postoperatively after one to two years. The primary surgical goals are the preservation of a clear graft and improvement of vision. Surgical outcomes are limited by donor-recipient junction mismatch, astigmatism, rejection, infection and wound dehiscence.

The femtosecond laser is a focusable, infrared laser capable of cutting tissue at various depths and in a range of patterns, and is currently being used to create corneal lamellar flaps in LASIK surgery. The laser parameters can be adjusted for submicron precision in cutting desired diameters, depths and shapes in the cornea, with minimal collateral injury. This technology is now capable of creating full-thickness corneal trephinations with customized locking edges at the graft-host junction between the donor and recipient corneas in Femtosecond Laser-Assisted Keratoplasty (FLAK). This approach may allow for better wound junction of the donor and recipient corneas, which in turn may also significantly reduce astigmatism, improve wound healing and visual recovery.

Although the femtosecond laser has been approved by the FDA for use in corneal transplants, it has not been compared to standard corneal transplant techniques. This pilot study will help us determine optimal femtosecond laser spot size, separation, fluency, and energy which result in the best graft-host fit. Surgical eligibility criteria, including preoperative diagnoses, as well as possible associated medical and ophthalmic conditions for the eventual multi-center study will be defined. Primary outcome measures, which include corneal refractive power measurements, serial endothelial-cell counts to assess endothelial survival and vision-specific quality of life surveys, will be evaluated. The specific aim is to investigate postoperative physiology and biomechanics after FLAK in human eyes. The significance is that FLAK presents corneal surgeons with an opportunity to avoid some problems of PKP and offers a safer and more precise approach to treating visually disabling diseases secondary to corneal opacification.

ELIGIBILITY:
Inclusion Criteria:

1. Corneal opacification.
2. Reduced ETDRS-measured, best corrected, distance visual acuity to 20/40 or worse.
3. Ability to participate in follow-up visits.
4. Signed, informed consent.

Exclusion Criteria:

1. Corneal opacification adequately dense to obscure visualization of iris.
2. ETDRS-measured, best-corrected, distance visual acuity of 20/30 or better.
3. Corneal thickness greater than 1200 µm at the 9 mm peripheral zone.
4. Severe corneal thinning including descemetocoele with impending corneal rupture.
5. Prior PKP or incisional surgery that may provide a potential space into which the gas produced by the procedure can escape.
6. Poor visual potential in the non-study eye (VA of 20/100 or less, without potential for improvement by the examining ophthalmologist's judgment).
7. History of glaucoma, including steroid response rise in intraocular pressure.
8. Active intraocular inflammation or infection.
9. Age 18 or younger.
10. Unable to return for scheduled follow-up examinations.
11. Other medical condition(s) that will likely prevent long term follow-up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Investigate postoperative physiology and biomechanics after Femtosecond Laser Assisted Keratoplasty in human eyes. | Preoperatively and 1day, 1week and 1, 3, 6, 12, 18 and 24 months post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Mian, MD, Principal Investigator — University of Michigan Kellogg Eye Center
Locations (1):
- Cornea Clinic, Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No